CLINICAL TRIAL: NCT02564614
Title: A Phase 1b, Proof of Mechanism, Open-label Study of RO7070179, a Hypoxia-inducible Factor 1a (HIF1A) mRNA Antagonist in Adult Subjects With Hepatocellular Carcinoma (HCC)
Brief Title: A Study of Hypoxia-inducible Factor 1a (HIF1A) Messenger Ribonucleic Acid (mRNA) Antagonist (RO7070179), to Demonstrate Proof-of-mechanism in Adult Participants With Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP29700
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

ARMS (1):
- RO7070179 (Experimental): Participants will receive RO7070179, 13 mg/kg/week, 2-hour IV infusion every week in a 6-week cycle, after two loading doses in Week 1 of Cycle 1 on Day 1 and Day 4. If a dose-limiting toxicity (DLT) occurs in more than 33% of participants at any time, the dose will be reduced to 10 mg/kg/week. The dose will be further reduced to 6 mg/kg/week if more than 33% of treated participants have a DLT.
  Interventions: Drug: RO7070179

INTERVENTIONS:
Drug: RO7070179 — RO7070179 (13 mg/kg/week) will be administered as 2-hour IV infusion.
  Other Names: SPC2968/EZN-2968

SUMMARY:
This open-label study will demonstrate proof-of-mechanism of HIF1A inhibition by a decrease of HIF1A mRNA after intravenous (IV) infusion of RO7070179 in participants with hepatocellular carcinoma (HCC) who have failed at least one line of systemic therapy. This will be a single arm study and all participants will receive RO7070179, 13 milligram per kilogram per week (mg/kg/week), 2-hour IV infusion on Days 1 and 4 during Week 1 of Cycle 1, followed by once weekly in 6 week cycle. Treatment with RO7070179 will be continued until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of >=18 years of age with the Eastern Cooperative Oncology Group (ECOG) performance status 0-1, Child-Pugh score of 5-7, and Life expectancy of 3 months or greater.
* Confirmed to have HCC as described by the American Association for the Study of Liver Disease (AASLD).
* Participants who have failed at least one line of systemic therapy for advanced stage HCC or participants who are ineligible or unable to tolerate the standard of care treatment.
* Have measurable or evaluable disease.
* Participants with normal major organ functions as defined by hemoglobin (HgB) >= 8.5 gram/decilitre (dL), absolute neutrophil count (ANC) >= 1000/microliter (mcL), platelet >= 60,000/micL, aspartate aminotransferase/alanine transaminase (AST/ALT) <= 3 x Upper Limit of Normal (ULN), total Bilirubin <= 2 x ULN, creatinine <= 2 x ULN.
* Willingness to undergo two tumor biopsies: before and after administration of RO7070179.

Exclusion Criteria:

* Concurrent serious medical illness that could potentially interfere with protocol compliance (such medical illness will not include hepatitis or cirrhosis, as the degree of liver impairment caused by these diseases are covered by other exclusion criteria).
* Active hepatitis B or C, but participants on stable medications for hepatitis B or C.
* Bleeding esophageal or gastric varices within 2 months before enrollment.
* Participants who need to take therapeutic anti-coagulation or anti-platelet therapy.
* Presence of ascites that preclude biopsy of liver lesions.
* History of unstable angina or myocardial infarction within 12 months prior to Day 1 or ischemic heart disease.
* Known HIV positive and positive screening pregnancy test or is breast-feeding.
* Female or male of reproductive capacity unwilling to use methods of contraception to prevent pregnancy during this study. Participants unwilling to use methods of contraception to prevent pregnancy for 6 months after the last dose of RO7070179 due to the potential for prolonged half-life of RO7070179 in the liver.
* Known, clinically suspected, or history of CNS tumor involvement.
* Prior chemotherapy, immunotherapy, investigational therapeutic agent, or other therapy used to treat HCC within 4 weeks before the first scheduled administration of RO7070179.
* Participants who have not recovered from any reversible side effects (except alopecia) to Grade 0 or 1 toxicity attributed to the administration of an investigational therapeutic agent, chemotherapy, immunotherapy, radiotherapy, or other agents previously used to treat the cancer.
* Any condition that, in the opinion of the investigator or the Sponsor, makes the patients unsuitable for the study.
* Inability to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-02; Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to Week 6 in HIF1A mRNA Level in Tumor Tissue | Pre-dose (baseline) and Week 6

SECONDARY OUTCOMES:
Change From Baseline to Week 6 in hypoxia-inducible factor 1a (HIF1A) Tumor Concentrations | Pre-dose (baseline) and Week 6
Change From Baseline to Week 6 in HIF2 Tumor Concentrations | Pre-dose (baseline) and Week 6
Change From Baseline to Week 6 in Vascular Endothelial Growth Factor (VEGF) Tumor Concentrations | Pre-dose (baseline) and Week 6
Change From Baseline to Week 6 in Erythropoietin (EPO) Tumor Concentrations | Pre-dose (baseline) and Week 6
Change From Baseline to Week 6 in Prolyl 4 Hydroxylase Tumor Concentrations | Pre-dose (baseline) and Week 6
Change From Baseline to Week 6 in CD34/von Willebrand factor (VWF) Tumor Concentrations | Pre-dose (baseline) and Week 6
Change in Blood Alpha-fetoprotein (AFP) Concentrations from Baseline | Week 1 and Week 4 for Cycle 1 and at Week 1 for subsequent treatment cycles
Time to Progression (TTP) According to Response Evaluation Criteria in Solid Tumors (RECIST) and modified RECIST (mRECIST) | Every 12 weeks upto 24 Months
Percentage of Participants With Complete Response (CR) and Partial Response (PR) According to RECIST and mRECIST | Every 12 weeks upto 24 Months
Duration of Response (DOR) According to RECIST and mRECIST | Every 12 weeks upto 24 Months
Progression Free Survival (PFS) According to RECIST and mRECIST | Every 12 weeks upto 24 Months
Overall Survival (OS) According to RECIST and mRECIST | Every 12 weeks upto 24 Months
Percentage of Participants With Tumor Growth According to RECIST and mRECIST | Every 12 weeks upto 24 Months
Maximum Observed Plasma Concentration (Cmax) | pre- and post-dose at Week 1, Week 6
Time to Reach Maximum Observed Plasma Concentration (Tmax) | pre- and post-dose at Week 1, Week 6
Area under the Concentration-Time Curve From Zero to 168 Hours [AUC (0-168 hours)] | pre- and post-dose at Week 1, Week 6
Plasma Decay Half-Life (t1/2) | pre- and post-dose at Week 1, Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (7):
  - Indiana University, Indianapolis, Indiana
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - NYU Langone Medical Center; Bellevue Hospital, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Ohio State University, Columbus, Ohio